CLINICAL TRIAL: NCT06014736
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Immunogenicity of XJ101 in Chinese Healthy Subjects
Brief Title: A Phase I Study of XJ101 in Chinese Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Starmab biologics（Shanghai）Co,.ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJ101-I
Record Dates: First submitted 2023-08-16; First posted 2023-08-28 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-01

CONDITIONS: Staphylococcus Aureus Bloodstream Infection
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XJ101 for Injection (Experimental): XJ101 via intravenous(IV).
  Interventions: Drug: XJ101 for Injection
- Placebo (Placebo Comparator): Placebo via intravenous(IV).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XJ101 for Injection — XJ101 is a recombinant humanized single domain antibody-Fc (human immunoglobulin G1 type) fusion protein.
  Arms: XJ101 for Injection
Drug: Placebo — Placebo contains only excipients.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-parallel intervention clinical study that will include approximately 38 healthy subjects based on inclusion and exclusion criteria. Subjects will be assigned to one of four different dosage cohorts. Subjects in each cohort will randomly be given experimental drug or a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 45 years at screening.
2. Male weight ≥ 50.0 kg, female weight ≥ 45.0 kg, and body mass index (BMI) within the range of 19.0 to 26.0 kg/m2 (including critical values).
3. The subjects have no pregnancy plan and voluntarily avoid pregnancy from signing the informed consent form until the end of the trail.
4. Healthy on the basis of physical examination and medical and surgical history and twelve-lead electrocardiogram (ECG) without clinically relevant abnormalities.
5. Written informed consent and any locally required authorization (eg, HIPAA) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

1. Subjects with any abnormalities of respiratory system, circulatory system, digestive system, nervous system, skeletal muscle system, blood and lymphatic system, immune system and endocrine system.
2. History of allergy to drugs or biological products.
3. Acute infection within 4 weeks prior to study entry.
4. Suffer from diseases caused by Staphylococcus aureus within one year, such as bacteremia, sepsis and pyemia.
5. Receipt of any standard vaccine within 4 weeks prior to investigational product dosing or plan to vaccinate during the study period.
6. Receipt of any major surgery within 3 months prior to the start of the trial, or have not recovered from surgery, or plan to have a surgical during the trial.
7. Those who cannot tolerate venipuncture, or have a history of injector and blood sickness, or are not suitable for venous blood collection.
8. Subjects with a history of drug abuse or drug use, or those with positive urine drug screening.
9. Blood donation or massive blood loss (> 200 mL) within three months prior to screening or plan to donate blood, receive blood transfusions, or use blood products during the trial period or within 1 month after the end of the trial.
10. Pregnant or lactating women.
11. Use of any prescription drugs, over-the-counter drugs, vitamin products or herbal medicines within 14 days prior to screening.
12. Smoke more than 5 cigarettes per day within three months prior to screening
13. Frequent drinkers in the three months before screening, i.e. those who drink more than or equal to 14 units of alcohol per week on average (1 unit=17.7 ml ethanol, 1 unit=354 ml beer with 5% alcohol, 44.25 ml spirits with 40% alcohol, or 147.5 ml wine with 12% alcohol), or those who do not agree to ban alcohol during the study period.
14. Evidence of infection with HBV, hepatitis C, HIV, or syphilis.
15. Positive alcohol breath test.
16. Subjects with special dietary requirements and cannot accept a unified diet.
17. Participation in other clinical trials within three months prior to enrollment or plan to participate in other clinical trials during this period.
18. Any other factors evaluated by investigators that patients cannot be enrolled.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Any adverse events that occurred among all subjects during the clinical trial, including clinical symptoms, vital signs or physical examination abnormalities, laboratory tests or 12-lead electrocardiogram abnormalities. | From the time of informed consent through 92 days post dose.

SECONDARY OUTCOMES:
Area Under the Serum Concentration Time Curve from Time Zero to Infinity (AUC [0-Infinity]) | From Day 1 through 92 days post dose.
Area Under the Serum Concentration Time Curve from Time Zero to Last Measurable Concentration (AUC [0-Last]) | From Day 1 through 92 days post dose.
Maximum Observed Serum Concentration (Cmax) | From Day 1 through 92 days post dose.
Terminal Phase Elimination Half-life (t1/2) | From Day 1 through 92 days post dose.
Elimination Rate Constant (Kel) | From Day 1 through 92 days post dose.
Mean Residence Time (MRT) | From Day 1 through 92 days post dose.
Apparent Serum Clearance (CL) | From Day 1 through 92 days post dose.
Apparent Volume of Distribution (Vd) | From Day 1 through 92 days post dose.
Percentage of Area Under the Serum Concentration Time Curve That Has Been Derived After Extrapolation (AUC_% Extrap) | From Day 1 through 92 days post dose.
Anti Drug Antibody (ADA) Assessments - Serum | From Day 1 through 92 days post dose.
  ADA responses to XJ101

CONTACTS AND LOCATIONS:
Overall Officials: Ding xueying, Study Director — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospita, Shanghai, Shanghai Municipality, China